CLINICAL TRIAL: NCT06216483
Title: Using EMR Data and AI to Develop a Passive Digital Marker to Predict Postoperative Delirium
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Sanjay Mohanty, Assistant Professor of Surgery, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 15767; K23AG071945 (NIH)
Record Dates: First submitted 2023-12-19; First posted 2024-01-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Delirium in Old Age

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No PDM Alert (Placebo Comparator): No PDM alert will be placed on subject's record
  Interventions: Other: PDM Alert
- PDM Alert (Experimental): PDM alert will be placed on subject's record
  Interventions: Other: PDM Alert

INTERVENTIONS:
Other: PDM Alert — passive digital marker (PDM) for postoperative delirium risk

SUMMARY:
This study will be a pilot randomized controlled trial that will determine the effect of an indicator of delirium risk, which will be delivered either via a paper form or via the electronic medical record, on (1)postoperative delirium incidence; and (2)the development of long term cognitive decline and dementia.

DETAILED DESCRIPTION:
Patients will be recruited from a large general, minimally invasive, colorectal, and oncologic, university-based surgical practice. English speaking individuals over the age of 65 with planned major abdominal surgery (encompassing abdominal wall, gastrointestinal and hepatobiliary procedures for benign and malignant diseases) will be screened for eligibility following an initial visit with their surgeon. Inclusion criteria will include a required inpatient stay for ≥ 24 hours following surgery and a scheduled preadmission testing and medical risk stratification visit with an internal medicine provider. Patients will be excluded if they have severe mental illness, hearing and visual impairment, alcohol intoxication or related delirium, central nervous disorder (e.g., stroke, traumatic brain injury), and pregnant or nursing status. Once enrolled, subjects will be randomized using a computer-generated scheme (permuted blocks of four and six) to the PDM or usual care, stratified according to type of surgery (hepatobiliary, gastrointestinal, abdominal wall).

ELIGIBILITY:
Inclusion Criteria:

65 years old Planned inpatient major surgery requiring inpatient stay ≥ 1 day

Exclusion Criteria:

* Baseline cognitive impairment or a diagnosis of Alzheimer's Disease/Alzheimer's Disease and Related Dementias (AD/ADRD)
* Alcohol or drug withdrawal
* Prisoner status
* Unable to communicate with research staff due to sensory impairments
* Not fluent in English
* Currently has a personal safety attendant

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Delirium incidence as measured by the 3D-CAM | Daily during post-operative inpatient hospitalization through post-operative day 7
  The number of subjects diagnosed with delirium via the 3D-CAM questionnaire will be measured. The 3D-CAM is a brief verbal assessment tool that can be used to test patients and study participants for delirium via the Confusion Assessment Method (CAM). The 3D-CAM assessment is scored as either delirium present or delirium not present. Participants will be evaluated daily during the acute post-operative phase of the study (Post-Operative Days 0-7).
Delirium incidence as measured by the CAM ICU | Daily during post-operative inpatient hospitalization through post-operative day 7
  The number of subjects diagnosed with delirium as assessed by the Confusion Assessment Method ICU will be measured. The CAM ICU is a tool used to assess delirium in adult ICU patients. CAM ICU scoring ranges from 0-7 with scores between 0-2 indicating no delirium, between 3-5 indicating mild to moderate delirium, and between 6-7 indicating severe delirium. Participants will be evaluated daily during the acute post-operative phase of the study (Post-Operative Days 0-7).
Delirium severity as measured by the CAM ICU | Daily during post-operative inpatient hospitalization through post-operative day 7
  Delirium severity will be assessed via the Confusion Assessment Method ICU, a tool used to assess delirium in adult ICU patients. The CAM ICU is a tool used to assess delirium in adult ICU patients. CAM ICU scoring ranges from 0-7 with scores between 0-2 indicating no delirium, between 3-5 indicating mild to moderate delirium, and between 6-7 indicating severe delirium. Participants will be evaluated daily during the acute post-operative phase of the study (Post-Operative Days 0-7).

SECONDARY OUTCOMES:
Inpatient falls | During post-operative inpatient hospitalization through post-operative day 7
  The number of inpatient falls will be compared between groups. This data will be extracted from the participants' Electronic Medical Record.
Restraint Use | During post-operative inpatient hospitalization through post-operative day 7
  Use of restraints will be compared between groups. This data will be extracted from the participants' Electronic Medical Record.
Sedative Use | During post-operative inpatient hospitalization through post-operative day 7
  Sedative use will be compared between groups. This data will be extracted from the participants' Electronic Medical Record.
Use of personal safety attendants | During post-operative inpatient hospitalization through post-operative day 7
  Personal safety attendant use will be compared between groups. This data will be extracted from the participants' Electronic Medical Record.
Provider Satisfaction | Within 2-6 weeks following participant discharge
  Provider satisfaction will be measured determined by a Simplified System Usability Scale (SSUS). The SSUS will be administered to providers within two weeks of the participant's discharge from the hospital, and providers will be asked to respond within 4 weeks of survey receipt. The SSUS yields a single number representing a composite measure of the overall usability of the system. Scores can range from 0 to 100, with higher scores indicating better usability.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Health University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No